CLINICAL TRIAL: NCT05654025
Title: Follow up Study on Visual Prognosis and Complications of Ectopia Lentis Lens
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KYPJ207
Record Dates: First submitted 2022-11-17; First posted 2022-12-16 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Ectopia Lentis; Dislocation, Lens
MeSH Terms: conditions — Ectopia Lentis; Lens Subluxation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-surgical group: Refractive change, ocular parameter changes, and prognosis without surgery: To evaluate the long-term changes in refractive state, ocular parameter, ocular development and visual prognosis in patients without congenital ectopia lentis surgery.
- Surgical group: Safety and efficacy of different congenital ectopia lentis surgeries: To compare the safety and efficacy of different congenital ectopia lentis surgeries, including phacoemulsification， phacoemulsification + Intraocular lens (IOL) implantation， phacoemulsification + IOL implantation + Capsular Tension Ring implantation or phacoemulsification + IOL implantation + transscleral fixation.

SUMMARY:
This is a single-centre, observational cohort study with the following objectives: Firstly, the investigators aim to evaluate the vision-related quality of life and mental health status in congenital ectopia lentis patients. Secondly, the investigators target to investigate the correlations between genotype and clinical phenotype in patients of congenital ectopia lentis. Thirdly, to explore the metabolic profiles in the aqueous humor (AH) of patients with congenital ectopia lentis. Lastly, this study aims to explore the longitudinal changes of ocular biological parameters and complications in patients with postoperative congenital ectopia lens in the Chinese population.

DETAILED DESCRIPTION:
Congenital ectopia lens is a rare ophthalmic disease that seriously harms the physical and mental health of patients. Surgery is the only definite treatment at present. However, the changes in vision-related quality of life, mental health status, ocular biological parameters postoperative congenital dislocation of lens have not been systematically studied in the Chinese population.

In this trial, the investigators aim to evaluate the vision-related quality of life and mental health status in congenital ectopia lentis patients, investigate the correlations between genotype and clinical phenotype in patients of congenital ectopia lentis, explore the metabolic profiles in the aqueous humor (AH) of patients with congenital ectopia lentis, and explore the longitudinal changes of ocular biological parameters and complications in patients with postoperative congenital ectopia lens in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital lens dislocation and age ≥ 3 years old.
* Agree to participate in this study with written informed consent from patients or legal guardians.

Exclusion Criteria:

* History of ophthalmic trauma or other ophthalmic surgeries.
* Combined with other ophthalmic diseases such as primary glaucoma, uveitis and corneal disease.
* Patients who could not cooperate in the examinations.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with congenital ectopia lentis at Zhongshan ophthalmic center.
Sampling Method: Non-Probability Sample
Enrollment: 604 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change of best corrected visual acuity | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation, 3 months, and 1, 2, 3 years postoperation
  Best corrected visual acuity (BCVA) is evaluated with an ETDRS chart at each visit.
Incidence of complications | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation, 3 months, and 1, 2, 3 years postoperation.
  Estimate the incidence of complications for both non-surgical group and surgical group.

SECONDARY OUTCOMES:
Change of axial length | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation, 3 months, and 1, 2, 3 years postoperation.
  Axial length will be evaluated with ZEISS IOLMaster 700 at each visit.
High order aberrations | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation, 3 months, and 1, 2, 3 years postoperation
  High order aberrations will be assessed with Nidek OPD-Scan III at each visit.
Central cornea endothelial cell loss | Preoperation, and 3 months, and 1, 2, 3 years postoperation
  Central cornea endothelial cell loss will be calculated with endokeratoscope in surgical group.
The state of zonules | Non-surgical group is assessed at first visit, and 1, 2, 3 years after enrollment. Surgical group will be assessed preoperation.
  The state of zonules will be assessed using ultrasound biomicroscopy.
Anterior chamber angle. | Non-surgical group is assessed at first visit, and 1, 2, 3 years after enrollment. Surgical group will be assessed preoperation, 3 months, and 1, 2, 3 years postoperation.
  Anterior chamber angle will be assessed using Tomey Casia 2 anterior segment optical coherence tomography (OCT).
Tilt and eccentricity of intraocular lens | 3 months, and 1, 2, 3 years postoperation
  Tilt and eccentricity of intraocular lens was evaluated with Pentacam in surgical group.
Intraocular pressure | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation, 3 months, and 1, 2, 3 years postoperation.
  Intraocular pressure with non-contact-tonometer at each visit.
Aortic root diameter | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation and 1, 2, 3 years postoperation
  Aortic root diameter will be measured using echocardiography.
Aortic Root (Sinuses of Valsalva) Z-score, adjusted by body-surface-area (Z-score) | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation and 1, 2, 3 years postoperation
  Z-Score will be calculated using the Marfan foundation's calculator (https://marfan.org/dx/zscore-children/). Normal Z-score range from -2 to 2. A dilated aortic root is defined as a Z-score ≥2.0. A larger Z-score is associated with an increased risk of aortic complications such as dissection, rupture, and valvular regurgitation.
Incidence of valvular heart disease | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation and 1, 2, 3 years postoperation
  The incidence of valvular heart disease (VHD) is defined as the ratio of patients diagnosed with VHD to the total number of patients enrolled.
Body mass index (BMI) | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation and 1, 2, 3 years postoperation.
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. The normal range for the Chinese population is 18.5 to 23.9. A high BMI can indicate high body fatness.
Metacarpophalangeal joint length | Non-surgical group is evaluated at first visit, and 1, 2, 3 years after enrollment. Surgical group is evaluated at preoperation and 1, 2, 3 years postoperation.
  Metacarpophalangeal joint length will be measured using palmar radiograph.
Choroidal thickness | Non-surgical group is evaluated at first visit and 3 years after enrollment. Surgical group is evaluated at preoperation and 3 years postoperation.
  Choroidal thickness will be measured with optical coherence tomography (OCT) images.
Choriocapillaris flow deficits | Non-surgical group is evaluated at first visit and 3 years after enrollment. Surgical group is evaluated at preoperation and 3 years postoperation.
  Choriocapillaris flow deficits will be measured with optical coherence tomography angiography (OCTA) images.
Genetic mutation state of patients | Preoperation
  Draw blood to detect the exact gene mutations in patients via whole-exome sequencing.
Vision-related quality of life | Non-surgical group is evaluated at first visit and 3 years after enrollment. Surgical group is evaluated at preoperation and 3 years postoperation.
  Vision-related quality of life will be assessed with the Pediatric Eye Questionnaire (PedEyeQ).

CONTACTS AND LOCATIONS:
Overall Officials: Danying Zheng, Principal Investigator — Guangdong Provincial Clinical Research Center for Ocular Diseases
Locations (1):
- Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual Science, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and results will be published in a peer-reviewed journal.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available on December 2027 for 10 years.
Access Criteria: Data are available upon reasonable request by contacting with the corresponding author.

REFERENCES:
- [Result] Kaur K, Gurnani B. Ectopia Lentis. 2023 Jun 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK578193/ PMID 35201721
- [Result] Lin J, Gong N, Cao Q, Zhou Y, Cai Y, Jin G, Young CA, Yang J, Wang Y, Zheng D. What hinders congenital ectopia lentis patients' follow-up visits? A qualitative study. BMJ Open. 2020 Mar 12;10(3):e030434. doi: 10.1136/bmjopen-2019-030434. PMID 32169922
- [Result] Guo D, Jin G, Zhou Y, Zhang X, Cao Q, Lian Z, Guo Y, Zheng D. Mutation spectrum and genotype-phenotype correlations in Chinese congenital ectopia lentis patients. Exp Eye Res. 2021 Jun;207:108570. doi: 10.1016/j.exer.2021.108570. Epub 2021 Apr 16. PMID 33844962
- [Result] Minsel WR, Bommert H, Pieritz R. [Relationship between speech--formal psychotherapeutic signs and results of client-centered discussion psychotherapy]. Z Klin Psychol Psychother. 1972;20(4):303-10. No abstract available. German. PMID 4662920
- [Result] Jin GM, Fan M, Cao QZ, Lin JX, Zhang YC, Lin JQ, Wang YY, Young CA, Zheng DY. Trends and characteristics of congenital ectopia lentis in China. Int J Ophthalmol. 2018 Sep 18;11(9):1545-1549. doi: 10.18240/ijo.2018.09.19. eCollection 2018. PMID 30225232
- [Result] Meng X, Cao X, Jia Y, Pan J, Du Y, Li X. Sutured Scleral Fixation of Posterior Chamber Intraocular Lens in Children under the Age of 9 with Congenital Ectopia Lentis. Ophthalmic Res. 2021;64(5):837-843. doi: 10.1159/000516324. Epub 2021 Jul 9. PMID 34247162
- [Result] Chen T, Chen J, Jin G, Zhang M, Chen Z, Zheng D, Jiang Y. Clinical Ocular Diagnostic Model of Marfan Syndrome in Patients With Congenital Ectopia Lentis by Pentacam AXL System. Transl Vis Sci Technol. 2021 Jun 1;10(7):3. doi: 10.1167/tvst.10.7.3. PMID 34061947
- [Result] Chen Z, Chen T, Zhang M, Chen J, Deng M, Zheng J, Lan LN, Jiang Y. Fibrillin-1 gene mutations in a Chinese cohort with congenital ectopia lentis: spectrum and genotype-phenotype analysis. Br J Ophthalmol. 2022 Dec;106(12):1655-1661. doi: 10.1136/bjophthalmol-2021-319084. Epub 2021 Jul 19. PMID 34281902
- [Result] Fuchs J, Rosenberg T. Congenital ectopia lentis. A Danish national survey. Acta Ophthalmol Scand. 1998 Feb;76(1):20-6. doi: 10.1034/j.1600-0420.1998.760105.x. PMID 9541430
- [Result] Zhang Y, Jin G, Young CA, Cao Q, Lin J, Lin J, Wang Y, Zheng D. Analysis of Corneal Astigmatism before Surgery in Chinese Congenital Ectopia Lentis Patients. Curr Eye Res. 2018 Aug;43(8):972-976. doi: 10.1080/02713683.2018.1470248. Epub 2018 May 23. PMID 29698085
- [Result] Liu L, Li X, Cao Q, Lian Z, Wu J, Jin G, Zheng D. A Modified Knotless Transscleral Intraocular Lens Fixation Technology for Congenital Ectopia Lentis. Ophthalmol Ther. 2023 Feb;12(1):99-110. doi: 10.1007/s40123-022-00586-9. Epub 2022 Oct 15. PMID 36243894
- [Result] Chen H, Ng KY, Li S, Jin G, Cao Q, Lian Z, Luo X, Ding X, Zheng D. CHARACTERISTICS OF THE FOVEAL MICROVASCULATURE IN CHILDREN WITH MARFAN SYNDROME: An Optical Coherence Tomography Angiography Study. Retina. 2022 Jan 1;42(1):138-151. doi: 10.1097/IAE.0000000000003272. PMID 34935768
- [Derived] Xu P, Ng K, Jin L, Young CA, Liu S, Liang X, Liu Z, Zhang X, Jin G, Zheng D. Visual prognosis and complications of congenital ectopia lentis: study protocol for a hospital-based cohort in Zhongshan Ophthalmic Center. BMJ Open. 2023 Jun 27;13(6):e072542. doi: 10.1136/bmjopen-2023-072542. PMID 37369426